CLINICAL TRIAL: NCT02803411
Title: Progression of AtheRosclerotic PlAque DetermIned by Computed TomoGraphic Angiography Imaging(PARADIGM)
Acronym: PARADIGM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Collaborators: Montreal Heart Institute (Other); Hospital da Luz, Portugal (Other); University of California, Los Angeles (Other); Centro Cardiologico Monzino (Other); University of British Columbia (Other); German Heart Institute (Other); National Institute of Cardiology, Laranjeiras, Brazil (Other Government); Weill Medical College of Cornell University (Other); Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Hyuk-Jae Chang, Professor, Yonsei University
Other Study IDs: 4-2016-0263
Record Dates: First submitted 2016-06-03; First posted 2016-06-17 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Coronary Heart Disease
Keywords: Coronary Heart Disease; Coronary Computed Tomography Angiography (CCTA); Coronary Atherosclerotic Plaque; coronary atherosclerosis
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To describe the natural history of the coronary atherosclerotic plaque development and progression over time by CCTA with demographic and laboratory data for refinement of risk stratification of patients referred for CCTA.

DETAILED DESCRIPTION:
All PARADIGM study patients underwent initial and follow-up CCTA based on order from their primary physician. Demographic data, targeted medical history, cardiovascular risk factors, and laboratory data was prospectively collected in electronic case report forms (eCRFs) at the time of the initial CCTA and at the time of follow-up CCTA.

ELIGIBILITY:
Inclusion Criteria:

* patients underwent two or more clinically indicated CCTA with 64-detector rows or greater for CAD evaluation
* patients underwent at least 2 year interval between the baseline and follow-up CCTA

Exclusion Criteria:

* poor image quality of CCTA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is patients with suspected or known CAD who had undergone serial CCTA by physician referral. Sites that had collected cohorts of CCTA patients with symptoms, risk factors, CCTA image data, and outcomes were invited to contribute data for a merged database. This sample includes patients with suspected or known CAD, and asymptomatic subjects undergoing CCTA for risk stratification to evaluate the significance of changes in CCTA findings in different clinical contexts.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2003-03; Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in plaque volume and composition detected by follow up CCTA | 2 years

SECONDARY OUTCOMES:
Cardiac mortality (yes or no) | 2 years
Myocardial infarction (yes or no) | 2 years
Unstable angina requiring hospitalization (yes or no) | 2 years
Revascularization (yes or no) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hyuk-Jae Chang, MD, PhD, Principal Investigator — Yonsei Univerity

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee SE, Chang HJ, Rizvi A, Hadamitzky M, Kim YJ, Conte E, Andreini D, Pontone G, Volpato V, Budoff MJ, Gottlieb I, Lee BK, Chun EJ, Cademartiri F, Maffei E, Marques H, Leipsic JA, Shin S, Choi JH, Chung N, Min JK. Rationale and design of the Progression of AtheRosclerotic PlAque DetermIned by Computed TomoGraphic Angiography IMaging (PARADIGM) registry: A comprehensive exploration of plaque progression and its impact on clinical outcomes from a multicenter serial coronary computed tomographic angiography study. Am Heart J. 2016 Dec;182:72-79. doi: 10.1016/j.ahj.2016.09.003. Epub 2016 Sep 22. PMID 27914502
- [Derived] Neglia D, Caselli C, Maffei E, Cademartiri F, Meloni A, Bossone E, Saba L, Lee SE, Sung JM, Andreini D, Al-Mallah MH, Budoff MJ, Chinnaiyan K, Choi JH, Chun EJ, Conte E, Gottlieb I, Hadamitzky M, Kim YJ, Lee BK, Leipsic JA, Marques H, de Araujo Goncalves P, Pontone G, Shin S, Stone PH, Samady H, Virmani R, Narula J, Shaw LJ, Bax JJ, Lin FY, Min JK, Chang HJ. Rapid Plaque Progression Is Independently Associated With Hyperglycemia and Low HDL Cholesterol in Patients With Stable Coronary Artery Disease: A PARADIGM Study. Circ Cardiovasc Imaging. 2024 Jul;17(7):e016481. doi: 10.1161/CIRCIMAGING.123.016481. Epub 2024 Jul 16. PMID 39012946
- [Derived] Park HB, Arsanjani R, Sung JM, Heo R, Lee BK, Lin FY, Hadamitzky M, Kim YJ, Conte E, Andreini D, Pontone G, Budoff MJ, Gottlieb I, Chun EJ, Cademartiri F, Maffei E, Marques H, Goncalves PA, Leipsic JA, Lee SE, Shin S, Choi JH, Virmani R, Samady H, Chinnaiyan K, Stone PH, Berman DS, Narula J, Shaw LJ, Bax JJ, Min JK, Chang HJ. Impact of statins based on high-risk plaque features on coronary plaque progression in mild stenosis lesions: results from the PARADIGM study. Eur Heart J Cardiovasc Imaging. 2023 Oct 27;24(11):1536-1543. doi: 10.1093/ehjci/jead110. PMID 37232393
- [Derived] Won KB, Lee BK, Lin FY, Hadamitzky M, Kim YJ, Sung JM, Conte E, Andreini D, Pontone G, Budoff MJ, Gottlieb I, Chun EJ, Cademartiri F, Maffei E, Marques H, de Araujo Goncalves P, Leipsic JA, Lee SE, Shin S, Choi JH, Virmani R, Samady H, Chinnaiyan K, Berman DS, Narula J, Shaw LJ, Bax JJ, Min JK, Chang HJ. Glycemic control is independently associated with rapid progression of coronary atherosclerosis in the absence of a baseline coronary plaque burden: a retrospective case-control study from the PARADIGM registry. Cardiovasc Diabetol. 2022 Nov 12;21(1):239. doi: 10.1186/s12933-022-01656-9. PMID 36371222
- [Derived] Won KB, Lee BK, Heo R, Park HB, Lin FY, Hadamitzky M, Kim YJ, Sung JM, Conte E, Andreini D, Pontone G, Budoff MJ, Gottlieb I, Chun EJ, Cademartiri F, Maffei E, Marques H, de Araujo Goncalves P, Leipsic JA, Lee SE, Shin S, Choi JH, Virmani R, Samady H, Chinnaiyan K, Berman DS, Narula J, Bax JJ, Min JK, Chang HJ. Longitudinal Quantitative Assessment of Coronary Atherosclerotic Plaque Burden Related to Serum Hemoglobin Levels. JACC Asia. 2022 Apr 12;2(3):311-319. doi: 10.1016/j.jacasi.2021.10.010. eCollection 2022 Jun. PMID 36338409
- [Derived] Lee SE, Sung JM, Andreini D, Al-Mallah MH, Budoff MJ, Cademartiri F, Chinnaiyan K, Choi JH, Chun EJ, Conte E, Gottlieb I, Hadamitzky M, Kim YJ, Lee BK, Leipsic JA, Maffei E, Marques H, de Araujo Goncalves P, Pontone G, Shin S, Kitslaar PH, Reiber JHC, Stone PH, Samady H, Virmani R, Narula J, Berman DS, Shaw LJ, Bax JJ, Lin FY, Min JK, Chang HJ. Association Between Changes in Perivascular Adipose Tissue Density and Plaque Progression. JACC Cardiovasc Imaging. 2022 Oct;15(10):1760-1767. doi: 10.1016/j.jcmg.2022.04.016. Epub 2022 Jun 15. PMID 36202455
- [Derived] Takagi H, Leipsic JA, Indraratna P, Gulsin G, Khasanova E, Tzimas G, Lin FY, Shaw LJ, Lee SE, Andreini D, Al-Mallah MH, Budoff MJ, Cademartiri F, Chinnaiyan K, Choi JH, Conte E, Marques H, de Araujo Goncalves P, Gottlieb I, Hadamitzky M, Maffei E, Pontone G, Shin S, Kim YJ, Lee BK, Chun EJ, Sung JM, Virmani R, Samady H, Stone PH, Berman DS, Narula J, Bax JJ, Chang HJ. Association of Tube Voltage With Plaque Composition on Coronary CT Angiography: Results From PARADIGM Registry. JACC Cardiovasc Imaging. 2021 Dec;14(12):2429-2440. doi: 10.1016/j.jcmg.2021.07.011. Epub 2021 Aug 18. PMID 34419398
- [Derived] Hwang D, Kim HJ, Lee SP, Lim S, Koo BK, Kim YJ, Kook W, Andreini D, Al-Mallah MH, Budoff MJ, Cademartiri F, Chinnaiyan K, Choi JH, Conte E, Marques H, de Araujo Goncalves P, Gottlieb I, Hadamitzky M, Leipsic JA, Maffei E, Pontone G, Raff GL, Shin S, Lee BK, Chun EJ, Sung JM, Lee SE, Berman DS, Lin FY, Virmani R, Samady H, Stone PH, Narula J, Bax JJ, Shaw LJ, Min JK, Chang HJ. Topological Data Analysis of Coronary Plaques Demonstrates the Natural History of Coronary Atherosclerosis. JACC Cardiovasc Imaging. 2021 Jul;14(7):1410-1421. doi: 10.1016/j.jcmg.2020.11.009. Epub 2021 Jan 13. PMID 33454260
- [Derived] Jin HY, Weir-McCall JR, Leipsic JA, Son JW, Sellers SL, Shao M, Blanke P, Ahmadi A, Hadamitzky M, Kim YJ, Conte E, Andreini D, Pontone G, Budoff MJ, Gottlieb I, Lee BK, Chun EJ, Cademartiri F, Maffei E, Marques H, de Araujo Goncalves P, Shin S, Choi JH, Virmani R, Samady H, Stone PH, Berman DS, Narula J, Shaw LJ, Bax JJ, Chinnaiyan K, Raff G, Al-Mallah MH, Lin FY, Min JK, Sung JM, Lee SE, Chang HJ. The Relationship Between Coronary Calcification and the Natural History of Coronary Artery Disease. JACC Cardiovasc Imaging. 2021 Jan;14(1):233-242. doi: 10.1016/j.jcmg.2020.08.036. Epub 2020 Nov 18. PMID 33221216
- [Derived] Kim M, Lee SP, Kwak S, Yang S, Kim YJ, Andreini D, Al-Mallah MH, Budoff MJ, Cademartiri F, Chinnaiyan K, Choi JH, Conte E, Marques H, de Araujo Goncalves P, Gottlieb I, Hadamitzky M, Leipsic JA, Maffei E, Pontone G, Raff GL, Shin S, Lee BK, Chun EJ, Sung JM, Lee SE, Berman DS, Lin FY, Virmani R, Samady H, Stone PH, Narula J, Bax JJ, Shaw LJ, Min JK, Chang HJ. Impact of age on coronary artery plaque progression and clinical outcome: A PARADIGM substudy. J Cardiovasc Comput Tomogr. 2021 May-Jun;15(3):232-239. doi: 10.1016/j.jcct.2020.09.009. Epub 2020 Oct 1. PMID 33032975
- [Derived] Lee SE, Sung JM, Andreini D, Al-Mallah MH, Budoff MJ, Cademartiri F, Chinnaiyan K, Choi JH, Chun EJ, Conte E, Gottlieb I, Hadamitzky M, Kim YJ, Lee BK, Leipsic JA, Maffei E, Marques H, de Araujo Goncalves P, Pontone G, Shin S, Stone PH, Samady H, Virmani R, Narula J, Berman DS, Shaw LJ, Bax JJ, Lin FY, Min JK, Chang HJ. Sex Differences in Compositional Plaque Volume Progression in Patients With Coronary Artery Disease. JACC Cardiovasc Imaging. 2020 Nov;13(11):2386-2396. doi: 10.1016/j.jcmg.2020.06.034. Epub 2020 Aug 19. PMID 32828763
- [Derived] Lee SE, Sung JM, Andreini D, Al-Mallah MH, Budoff MJ, Cademartiri F, Chinnaiyan K, Choi JH, Chun EJ, Conte E, Gottlieb I, Hadamitzky M, Kim YJ, Lee BK, Leipsic JA, Maffei E, Marques H, de Araujo Goncalves P, Pontone G, Shin S, Stone PH, Samady H, Virmani R, Narula J, Berman DS, Shaw LJ, Bax JJ, Lin FY, Min JK, Chang HJ. Per-lesion versus per-patient analysis of coronary artery disease in predicting the development of obstructive lesions: the Progression of AtheRosclerotic PlAque DetermIned by Computed TmoGraphic Angiography Imaging (PARADIGM) study. Int J Cardiovasc Imaging. 2020 Dec;36(12):2357-2364. doi: 10.1007/s10554-020-01960-z. Epub 2020 Aug 10. PMID 32779077
- [Derived] Won KB, Lee BK, Park HB, Heo R, Lee SE, Rizvi A, Lin FY, Kumar A, Hadamitzky M, Kim YJ, Sung JM, Conte E, Andreini D, Pontone G, Budoff MJ, Gottlieb I, Chun EJ, Cademartiri F, Maffei E, Marques H, de Araujo Goncalves P, Leipsic JA, Shin S, Choi JH, Virmani R, Samady H, Chinnaiyan K, Raff GL, Stone PH, Berman DS, Narula J, Shaw LJ, Bax JJ, Min JK, Chang HJ. Quantitative assessment of coronary plaque volume change related to triglyceride glucose index: The Progression of AtheRosclerotic PlAque DetermIned by Computed TomoGraphic Angiography IMaging (PARADIGM) registry. Cardiovasc Diabetol. 2020 Jul 18;19(1):113. doi: 10.1186/s12933-020-01081-w. PMID 32682451
- [Derived] Lee SE, Sung JM, Andreini D, Al-Mallah MH, Budoff MJ, Cademartiri F, Chinnaiyan K, Choi JH, Chun EJ, Conte E, Gottlieb I, Hadamitzky M, Kim YJ, Lee BK, Leipsic JA, Maffei E, Marques H, de Araujo Goncalves P, Pontone G, Raff GL, Shin S, Stone PH, Samady H, Virmani R, Narula J, Berman DS, Shaw LJ, Bax JJ, Lin FY, Min JK, Chang HJ. Differences in Progression to Obstructive Lesions per High-Risk Plaque Features and Plaque Volumes With CCTA. JACC Cardiovasc Imaging. 2020 Jun;13(6):1409-1417. doi: 10.1016/j.jcmg.2019.09.011. Epub 2019 Nov 13. PMID 31734214
- [Derived] Won KB, Lee SE, Lee BK, Park HB, Heo R, Rizvi A, Hadamitzky M, Kim YJ, Sung JM, Conte E, Andreini D, Pontone G, Budoff MJ, Gottlieb I, Chun EJ, Cademartiri F, Maffei E, Marques H, Leipsic JA, Shin S, Choi JH, Virmani R, Samady H, Stone PH, Berman DS, Narula J, Shaw LJ, Bax JJ, Min JK, Chang HJ. Longitudinal quantitative assessment of coronary plaque progression related to body mass index using serial coronary computed tomography angiography. Eur Heart J Cardiovasc Imaging. 2019 May 1;20(5):591-599. doi: 10.1093/ehjci/jey192. PMID 30657884
- [Derived] Won KB, Lee SE, Lee BK, Park HB, Heo R, Rizvi A, Lin FY, Kumar A, Hadamitzky M, Kim YJ, Sung JM, Conte E, Andreini D, Pontone G, Budoff MJ, Gottlieb I, Chun EJ, Cademartiri F, Maffei E, Marques H, Leipsic JA, Shin S, Choi JH, Virmani R, Samady H, Chinnaiyan K, Raff GL, Stone PH, Berman DS, Narula J, Shaw LJ, Bax JJ, Min JK, Chang HJ. Longitudinal assessment of coronary plaque volume change related to glycemic status using serial coronary computed tomography angiography: A PARADIGM (Progression of AtheRosclerotic PlAque DetermIned by Computed TomoGraphic Angiography Imaging) substudy. J Cardiovasc Comput Tomogr. 2019 Mar-Apr;13(2):142-147. doi: 10.1016/j.jcct.2018.12.002. Epub 2018 Dec 17. PMID 30580992
- [Derived] Lee SE, Sung JM, Rizvi A, Lin FY, Kumar A, Hadamitzky M, Kim YJ, Conte E, Andreini D, Pontone G, Budoff MJ, Gottlieb I, Lee BK, Chun EJ, Cademartiri F, Maffei E, Marques H, Leipsic JA, Shin S, Hyun Choi J, Chinnaiyan K, Raff G, Virmani R, Samady H, Stone PH, Berman DS, Narula J, Shaw LJ, Bax JJ, Min JK, Chang HJ. Quantification of Coronary Atherosclerosis in the Assessment of Coronary Artery Disease. Circ Cardiovasc Imaging. 2018 Jul;11(7):e007562. doi: 10.1161/CIRCIMAGING.117.007562. PMID 30012825
- [Derived] Lee SE, Chang HJ, Sung JM, Park HB, Heo R, Rizvi A, Lin FY, Kumar A, Hadamitzky M, Kim YJ, Conte E, Andreini D, Pontone G, Budoff MJ, Gottlieb I, Lee BK, Chun EJ, Cademartiri F, Maffei E, Marques H, Leipsic JA, Shin S, Choi JH, Chinnaiyan K, Raff G, Virmani R, Samady H, Stone PH, Berman DS, Narula J, Shaw LJ, Bax JJ, Min JK. Effects of Statins on Coronary Atherosclerotic Plaques: The PARADIGM Study. JACC Cardiovasc Imaging. 2018 Oct;11(10):1475-1484. doi: 10.1016/j.jcmg.2018.04.015. Epub 2018 Jun 13. PMID 29909109